CLINICAL TRIAL: NCT02915224
Title: A Multicenter, Single Arm, Non-Interventional, Observational Study of Obinutuzumab to Evaluate Efficacy, Safety and Cost of Disease Management in Patients With Chronic Lymphocytic Leukemia and Comorbidities in Greece
Brief Title: A Study of Obinutuzumab Evaluating Efficacy, Safety and Cost of Disease Management in Participants With Chronic Lymphocytic Leukemia and Comorbidities
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30133
Record Dates: First submitted 2016-09-23; First posted 2016-09-26 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Chlorambucil; obinutuzumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Obinutuzumab: Participants will receive obinutuzumab as per Summary of Product Characteristics in daily practice along with chlorambucil for 24 months.
  Interventions: Drug: Chlorambucil; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Chlorambucil — Participants will receive chlorambucil as per summary of product characteristics in daily practice. Protocol does not specify any dosage.
Drug: Obinutuzumab — Participants will receive obinutuzumab as per summary of product characteristics in daily practice. Protocol does not specify any dosage.
  Other Names: Gazyvaro®

SUMMARY:
This multicenter, single arm, non-interventional, observational study will evaluate the efficacy and safety of obinutuzumab in daily clinical practice in participants with chronic lymphocytic leukemia (CLL). The study will also assess cost of disease management. The total length of the study is 42 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with untreated CLL and comorbidities, for which the physician has already decided to use obinutuzumab in association with chlorambucil

Exclusion Criteria:

* Participation in another clinical trial during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving obinutuzumab for CLL and comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS)\n | From screening every 6 months to Month 18 until disease progression (up to 24 months)

SECONDARY OUTCOMES:
Overall Survival (OS) | From screening every 6 months to Month 18 until disease progression (up to 24 months)
Percentage of Participants With Overall Response as Assessed by Investigator | From screening every 6 months to Month 18 until disease progression (up to 24 months)
Time to Response | From screening every 6 months to Month 18 until disease progression (up to 24 months)
Percentage of Participants With Best Overall Response as Assessed by Investigator | From screening every 6 months to Month 18 until disease progression (up to 24 months)
Time to Next Treatment, Defined as the Time Between the Date of Enrollment and First Intake of New Anti-Leukemic Therapy | Baseline up to 24 months
Duration of Response | From screening every 6 months to Month 18 until disease progression (up to 24 months)
Percentage of Participants With Protocol Defined Adverse Events of Special Interest | Baseline up to 24 months
Percentage of Participants With Protocol Defined Adverse Events of Particular Interest | Baseline up to 24 months
Percentage of Participants With Dose Delays/Discontinuations | Baseline up to 24 months
Percentage of Participants With Hematological Toxicities | Baseline up to 24 Months
Percentage of Participants With Non-hematological Toxicities | Baseline up to 24 months
Number of Hospital Admissions | Baseline up to 24 months
Number of Physician Visits | Baseline up to 24 months
Number of Diagnostic and Lab Exams | Baseline up to 24 months
Number of Medical Procedures (Blood Transfusions, Bone Marrow, or Stem Cell Transplantation) | Baseline up to 24 months
Costs of Treatment With Obinutuzumab | Baseline up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Greece (11):
  - University General Hospital of Alexandroupolis; Haemotology, Alexandroup
  - Laiko General Hospital of Athens; A Propedeutical Clinic of Internal Medicine, Athens
  - Laiko General Hospital; Hematology Clinic, Athens
  - General Hospital G. Gennimatas; Hematology Dept., Athens
  - Attiko Hospital; Haematology Clinic, Athens
  - Periph. University General Hospital of Heraklion; Hematology, Heraklion
  - University Hospital of Larissa; Hematology Dept., Larissa
  - University General Hospital of Patra; Internal Medicine Clinic - Hematology Department, Pátrai
  - Metaxa Hospital; Hematology Clinic, Piraeus
  - AXEPA Pathology Section; A Pathology Clinic, Thessaloniki
  - General Hospital G. Papanikolaou; Hematology, BMT Unit, Thessaloniki